CLINICAL TRIAL: NCT02684604
Title: Anti-Helicobacter Pylori Antibodies (IgG) in Serum of Women With Unexplained Infertility
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud Riad, Lecturer of obstetrics and gynecology, Ain Shams Maternity Hospital
Other Study IDs: unexplained infertility
Record Dates: First submitted 2016-02-08; First posted 2016-02-18 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- unexplained infertility patients: 44 patients diagnosed to have unexplained infertility
- Fertile women: 44 fertile women

SUMMARY:
Prevalence of anti-H.pylori IgG in serum of women with unexplained infertility and comparing that with it's prevalence in fertile women.

DETAILED DESCRIPTION:
Unexplained infertility was diagnosed according to standard World Health Organization (WHO) criteria. All women in the study had hormonal assessment to evaluate their ovulatory cycles, thyroid function, circulating prolactin and androgen levels. The ovarian reserve was checked by measurement of serum FSH and an antral follicle count on the third day of the menstrual cycle. Screening for infertility also included transvaginal ultrasound and hysterosalpingography, to exclude possible uterine malformations or pathologies, and to assess the patency of the fallopian tubes. Male factor infertility was excluded in all couples, according to standard WHO semen analysis.

Following admission, all patients underwent complete clinical examination and detailed medical history was obtained.

A venous sample was collected to test serum for HP IgG seropositivity by enzyme linked immunoassay for HELICOBACTOR PYLORI IgG (ENZYME IMMUNOASSAY TEST KIT).

ELIGIBILITY:
Inclusion Criteria:

1. regular cycles.
2. normal thyroid function, prolactin and androgen levels.
3. normal semen analysis of the partner.
4. normal hysterosalpingography.
5. normal transvaginal ultrasound examination.

Exclusion Criteria:

1. possible uterine malformations or pathologies.
2. presence of infections, including hepatitis, human immunodeﬁciency virus (HIV), TORCH, Chlamydia trachomatis and Mycoplasma.
3. presence of anti-sperm antibodies in serum.
4. Male factor infertility.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female healthy participants who attend the outpatient clinic
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unexplained Infertility Patients | Fertile Women
Started | 44 | 44
Completed | 44 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Normally distributed numerical variables were presented as mean and SD, and skewed variables as median and interquartile range. Comparison of normally distributed numerical data was done using the unpaired t test. Skewed data were compared using the Mann-Whitney U test. Ordinal data were compared using the chi-squared test for trend.
Groups:
- Total: Total of all reporting groups
Arm/Group | Unexplained Infertility Patients | Fertile Women | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (5.4) | 27.8 (4.9) | 28.06 (5.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 0 | 0 | 0
parity [Number; unit: participants]
  nullipara | 41 | 0 | 41
  para 1 | 2 | 13 | 15
  para 2 | 1 | 20 | 21
  para 3 | 0 | 10 | 10
  para 4 | 0 | 1 | 1
type of infertility [Number; unit: participants]
  no infertility | 0 | 44 | 44
  primary infertility | 41 | 0 | 41
  secondary infertility | 3 | 0 | 3
serum FSH level [Mean (Standard Deviation); unit: international unit per litre] | 6.85 (2.17) | 4.21 (1.85) | 5.53 (3.12)
serum LH level [Mean (Standard Deviation); unit: international unit per litre] | 5.43 (2.69) | 4.41 (3.21) | 4.92 (2.11)
serum prolactin level [Mean (Standard Deviation); unit: nanogram per millilitre] | 8.23 (3.39) | 9.21 (4.91) | 8.72 (3.45)
serum estradiole level [Mean (Standard Deviation); unit: picogram per millilitre] | 47.56 (16.55) | 34.52 (12.41) | 41.04 (14.02)
serum progesterone level [Mean (Standard Deviation); unit: nanogram per millilitre] | 14.09 (4.91) | 15.01 (5.21) | 14.55 (5.52)

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Helicobacter Pylori IgG Assay in Serum
Description: calculation of quantitative Helicobacter pylori IgG assay in serum
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: arbitrary unit per millilitre
Arm/Group | Unexplained Infertility Patients | Fertile Women
Number analyzed (Participants) | 44 | 44
arbitrary unit per millilitre | 70 [7.5 to 70] | 70 [70 to 70]
Statistical Analysis 1: Comparison: Unexplained Infertility Patients vs Fertile Women; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Unexplained Infertility Patients | Fertile Women
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No